CLINICAL TRIAL: NCT04231149
Title: Explorative Clinical Study Investigating the Performance and Acceptance of New Intermittent Catheters in Healthy Volunteers
Brief Title: Explorative Clinical Study on the Performance and Acceptance of New Intermittent Catheters in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CP290
Record Dates: First submitted 2019-05-28; First posted 2020-01-18 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Compliance, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product 2 (Experimental): Test catheter 2
  Interventions: Device: Test product 3; Device: Comparator
- Test product 3 (Experimental): Test catheter 3
  Interventions: Device: Test product 2; Device: Comparator
- Comparator (Active Comparator): SpeediCath Flex
  Interventions: Device: Test product 2; Device: Test product 3

INTERVENTIONS:
Device: Test product 2 — Test catheter 2
  Arms: Comparator; Test product 3
Device: Test product 3 — Test catheter 3
  Arms: Comparator; Test product 2
Device: Comparator — SpeediCath Flex
  Arms: Test product 2; Test product 3

SUMMARY:
Performance and acceptance of new intermittent catheters tested in healthy volunteers

DETAILED DESCRIPTION:
This study is a single blinded, randomised, crossover study. The study period consists of an information visit, an inclusion visit, three test visits and a termination visit.

Two prototypes of intermittent catheters (Test product 2 and 3) compared to the standard catheter SpeediCath® Flex (Comparator).

In the investigation ten subjects will be included. The subjects will be catheterised once per visit. The subjects will be catheterised with the two test catheters and comparator in a randomised order. The order of the catheterisations will be randomised to prevent bias.

During the test visits the primary, secondary and explorative endpoints will be registered.

Subjects will be asked to participate in an interview in continuation of their last visit (Test Visit 3). The interviews will be performed by a Coloplast representative asking questions related to their experience with the catheter.

The subjects must sign a separate consent form for this purpose and can participate in the investigation without participating in the interview. In addition, subjects will be asked for consent to tape recording and filming during the interviews, but can participate in interviews without this.

In addition, a Coloplast representative will interview the Investigator and her representatives after LPO with questions related to their experience with the catheters.

The investigation is planned to be conducted in August 2018-Januar 2019. The visit window will be minimum five days between the visits (catheterisations), to ensure time for healing of any potential urethral trauma. However, the maximum time between visits should be adjusted to ensure the subject is terminated before LPO.

No biobank will be established for this investigation. All urine samples in the clinical investigation (for evaluating in- and exclusion criteria and for evaluating end points) will be destructed immediately after analysis.

ELIGIBILITY:
Inclusion Criteria:

Has given written informed consent and signed letter of authority Is at least 18 years of age and has full legal capacity Is a male Willing to comply without using analgetica up to 24 hours prior to catheterisation visits

Exclusion Criteria:

Has a previous history of genitourinary disease including congenital abnormalities and surgical procedures performed in the urinary tract Has symptoms of urinary tract infections (frequent urination, stinging and pain at urination) Are participating in any other clinical investigation related to urinary tract system during this investigation (inclusion to termination) Known hypersensitivity toward any of the test products

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects need a penis for male urinary catheter use
Enrollment: 9 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects were screened for eligibility
Pre-assignment Details: 9 out of 10 were randomized. The one not randomized did not meet the inclusion criteria.
Groups:
- Test Product 2, Then Test Product 3, Then SpeediCath Flex: Participants were first catheterized with Test Product 2 at Visit 1. After a washout period of minimum 5 days, they were then catheterized with Test Product 3 at Visit 2. After a washout period of minimum 5 days again, they were then catheterized with SpeediCath Flex.
- Test Product 3, Then Test Product 2, Then SpeediCath Flex: Participants were first catheterized with Test Product 3 at Visit 1. After a washout period of minimum 5 days, they were then catheterized with Test Product 2 at Visit 2. After a washout period of minimum 5 days again, they were then catheterized with SpeediCath Flex.
- SpeediCath Flex, Then Test Product 2, Then Test Product 3: Participants were first catheterized with SpeediCath Flex at Visit 1. After a washout period of minimum 5 days, they were then catheterized with Test Product 2 at Visit 2. After a washout period of minimum 5 days again, they were then catheterized with Test Product 3.
- Test Product 2, Then SpeediCath Flex, Then Test Product 3: Participants were first catheterized with Test Product 2 at Visit 1. After a washout period of minimum 5 days, they were then catheterized with SpeediCath Flex at Visit 2. After a washout period of minimum 5 days again, they were then catheterized with Test Product 3.
- Test Product 3, Then SpeediCath Flex, Then Test Product 2: Participants were first catheterized with Test Product 3 at Visit 1. After a washout period of minimum 5 days, they were then catheterized with SpeediCath Flex at Visit 2. After a washout period of minimum 5 days again, they were then catheterized with Test Product 2.
Period: First Intervention (Visit 1)
Arm/Group | Test Product 2, Then Test Product 3, Then SpeediCath Flex | Test Product 3, Then Test Product 2, Then SpeediCath Flex | SpeediCath Flex, Then Test Product 2, Then Test Product 3 | Test Product 2, Then SpeediCath Flex, Then Test Product 3 | Test Product 3, Then SpeediCath Flex, Then Test Product 2
Started | 2 | 3 | 2 | 1 | 1
Completed | 2 | 3 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout (Minimum 5 Days)
Arm/Group | Test Product 2, Then Test Product 3, Then SpeediCath Flex | Test Product 3, Then Test Product 2, Then SpeediCath Flex | SpeediCath Flex, Then Test Product 2, Then Test Product 3 | Test Product 2, Then SpeediCath Flex, Then Test Product 3 | Test Product 3, Then SpeediCath Flex, Then Test Product 2
Started | 2 | 3 | 2 | 1 | 1
Completed | 2 | 3 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (Visit 2)
Arm/Group | Test Product 2, Then Test Product 3, Then SpeediCath Flex | Test Product 3, Then Test Product 2, Then SpeediCath Flex | SpeediCath Flex, Then Test Product 2, Then Test Product 3 | Test Product 2, Then SpeediCath Flex, Then Test Product 3 | Test Product 3, Then SpeediCath Flex, Then Test Product 2
Started | 2 | 3 | 2 | 1 | 1
Completed | 2 | 3 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout (Minimum 5 Days)
Arm/Group | Test Product 2, Then Test Product 3, Then SpeediCath Flex | Test Product 3, Then Test Product 2, Then SpeediCath Flex | SpeediCath Flex, Then Test Product 2, Then Test Product 3 | Test Product 2, Then SpeediCath Flex, Then Test Product 3 | Test Product 3, Then SpeediCath Flex, Then Test Product 2
Started | 2 | 3 | 2 | 1 | 1
Completed | 2 | 2 | 2 | 1 | 1
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Third Intervention (Visit 3)
Arm/Group | Test Product 2, Then Test Product 3, Then SpeediCath Flex | Test Product 3, Then Test Product 2, Then SpeediCath Flex | SpeediCath Flex, Then Test Product 2, Then Test Product 3 | Test Product 2, Then SpeediCath Flex, Then Test Product 3 | Test Product 3, Then SpeediCath Flex, Then Test Product 2
Started | 2 | 2 | 2 | 1 | 1
Completed | 2 | 2 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: The baseline measures include all study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 35.9 [20 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 9
Number of Participants with Hematuria at baseline [Count of Participants; unit: Participants] — Count of number of participants with hematuria at baseline
  Participants | 0

OUTCOME MEASURES:

1. Primary Outcome: Urine Flow Rate
Description: On day of study visits 1-5 rate of urine flow through catheter measured in mL/s
Time Frame: 2 hour
Measure: Mean (Full Range); unit: mL per second
Arm/Group | Test Product 2 | Test Product 3 | Comparator
Number analyzed (Participants) | 9 | 9 | 8
mL per second | 5.43 [3 to 8] | 5.47 [4 to 7] | 2.88 [2 to 4]

2. Secondary Outcome: Post-void Residual Urine
Description: On day of study visits 1-5 rate volume of urine left in the bladder post catheterisation (in mL)
Time Frame: 2 hour
Measure: Mean (Full Range); unit: mL
Arm/Group | Test Product 2 | Test Product 3 | Comparator
Number analyzed (Participants) | 9 | 9 | 8
mL | 38.33 [7 to 97] | 34.63 [12 to 88] | 27.75 [7 to 64]

3. Secondary Outcome: Number of Participants With Hematuria
Description: On day of study visits 1-5 blood in urine post catheterisation (measured as yes/no to blood in urine)
Time Frame: 2 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 2 | Test Product 3 | Comparator
Number analyzed (Participants) | 9 | 9 | 8
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Two hours on days of study visits 1-6 and termination visit
Arm/Group | Test Product 2 | Test Product 3 | Comparator
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT04231149/Prot_SAP_000.pdf